CLINICAL TRIAL: NCT04061057
Title: Effect of Perioperative Intravenous Lidocaine Infusion on Postoperative Recovery in Patients Undergoing Arthroscopic Rotator Cuff Repair Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2018-0033
Record Dates: First submitted 2019-08-12; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV lidocaine (Experimental): Perioperative IV lidocaine infusion
  Interventions: Drug: Lidocaine
- Normal saline (Placebo Comparator): Perioperative IV normal saline infusion
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — Drug: 1. Lidocaine Intravenous lidocaine bolus of 1.5mg/kg immediately after anesthesia induction followed by infusion at 2.0mg/kg/hr up to 1 hr after end of surgery.
  2. Fentanyl IV infusion via PCA (patient controlled analgesia) machine of fentanyl 10 μg/ml, ramosetron 0.3 mg, normal saline, total 100 ml, infusion rate 1 ml/hr, 1 ml bolus and lockout time 7 min.
  Arms: IV lidocaine
Drug: Normal saline — Drug: 1. Normal saline Intravenous normal saline bolus of immediately after anesthesia induction followed by infusion up to 1 hr after end of surgery. Volume of normal saline is equal to lidocaine.
  2. Fentanyl IV infusion via PCA (patient controlled analgesia) machine of fentanyl 10 μg/ml, ramosetron 0.3 mg, normal saline, total 100 ml, infusion rate 1 ml/hr, 1 ml bolus and lockout time 7 min.
  Arms: Normal saline

SUMMARY:
Arthroscopic rotator cuff repair is a commonly performed procedure but is known to cause significant postoperative pain. Effective analgesia after rotator cuff repair is crucial in improving the well-being of the patient but also to ensure long-term rehabilitation. The most commonly used analgesic for acute postoperative pain is opioids. However, the use of opioids is accompanied by several side effects which include but are not limited to nausea/vomiting, urinary retention, itching sensation and sometimes dizziness, respiratory depression and hypotension in higher doses. As of late, many efforts are aimed toward decreasing the use of opioids by using multimodal analgesia. Among such methods, intravenous lidocaine has been reported to be effective, safe and economic in various procedures. However, the existing evidence is mostly focused on laparoscopic procedures. The present study aims to find whether perioperative infusion of lidocaine is able to decrease opioid requirements after surgery and also improve postoperative pain compared to placebo in patients undergoing arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class 1-3 adults over 19 years scheduled for elective arthroscopic rotator cuff repair

Exclusion Criteria:

1. Known allergies to lidocaine or propofol
2. Cardia arrhythmia
3. History of epilepsy or seizures
4. Liver/kidney failure
5. History of recent strong opioid use

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Fentanyl requirement using IV PCA | 24hours after surgery
  Dose of fentanyl infused via IV PCA machine during first 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kim SJ, Choi YS, Chun YM, Kim HJ, Han C, Shin S. Perioperative Intravenous Lidocaine Infusion on Postoperative Recovery in Patients Undergoing Arthroscopic Rotator Cuff Repair Under General Anesthesia: A Randomized Controlled Trial. Clin J Pain. 2021 Oct 12;38(1):1-7. doi: 10.1097/AJP.0000000000000995. PMID 34636752